CLINICAL TRIAL: NCT05268484
Title: Improving Anticipatory and Compensatory Postural Responses to Avoid Falls After TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1072-19
Record Dates: First submitted 2022-02-25; First posted 2022-03-07 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- TBI Intervention Group (Experimental): Participants will participate in 16 anticipatory postural adjustments (APA) and compensatory postural adjustments (CPA) training sessions using the Neurocom Balance Platform. Each session will last for 1 hour. During the APA portion, a visual cue on the front screen in the form of a countdown timer showing the remaining seconds to the onset of the upcoming perturbation. This information will allow an opportunity for the participant to adjust their posture to handle the upcoming perturbation in the best possible way and also train them to anticipate upcoming disturbances and execute corrective motor outputs. This will ensure the generation of APA in a consistent and repetitive manner. In CPA, after a 5 second pause, the platform will oscillate at 1 Hz, with a constant amplitude, in the anterior-posterior direction for 50 seconds, followed by an additional 5 second quiet period. The participant will wear a safety harness at all times and a spotter will be present at all times.
  Interventions: Device: Perturbation-based Training with visual cues using Neurocom
- TBI Control Group (No Intervention): No intervention is provided
- Healthy Control (No Intervention): No intervention is provided

INTERVENTIONS:
Device: Perturbation-based Training with visual cues using Neurocom — Participants will participate in 16 anticipatory postural adjustments (APA) and compensatory postural adjustments (CPA) training sessions using the Neurocom Balance Platform. Each session will last for 1 hour. During the APA portion, a visual cue on the front screen in the form of a countdown timer showing the remaining seconds to the onset of the upcoming perturbation. This information will allow an opportunity for the participant to adjust their posture to handle the upcoming perturbation in the best possible way and also train them to anticipate upcoming disturbances and execute corrective motor outputs. This will ensure the generation of APA in a consistent and repetitive manner. In CPA, after a 5 second pause, the platform will oscillate at 1 Hz, with a constant amplitude, in the anterior-posterior direction for 50 seconds, followed by an additional 5 second quiet period. The participant will wear a safety harness at all times and a spotter will be present at all times.
  Other Names: Perturbation-based Training with visual cues (PBTvc)
  Arms: TBI Intervention Group

SUMMARY:
The purpose of this study is to assess a balance training program to see if it can be helpful to avoid falls in people who have had traumatic brain injuries (TBIs).

The study will include 3 groups: TBI Intervention group , TBI Control Group, and healthy control group.

TBI Intervention group - These individuals will participate in 16 anticipatory postural adjustments (APA) and compensatory postural adjustments (CPA) training sessions using the Neurocom Balance Platform. Each session will last for 1 hour. During the APA portion, participants will be provided with a visual cue on the front screen in the form of a countdown timer showing the remaining seconds to the onset of the upcoming perturbation. This information will allow an opportunity for the participant to adjust their posture to handle the upcoming perturbation in the best possible way and also train them to anticipate upcoming disturbances and execute corrective motor outputs. In CPA, after a 5 second pause, the platform will oscillate at 1 Hz, with a constant amplitude, in the anterior-posterior direction for 50 seconds, followed by an additional 5 second quiet period. The participant will wear a safety harness at all times and a spotter will be present at all times.

TBI Control Group- They do not receive any intervention. healthy control group- They do not receive any intervention.

All three groups will participate in two data collection sessions: Baseline and follow-up.

At baseline and follow-up, we will collect functional, clinical, biomechanical, and physiological metrics.

During training and data collection, a spotter will be present at all times to prevent falls and participants will be allowed as much rest as needed by them..

ELIGIBILITY:
INCLUSION CRITERIA FOR TRAUMATIC BRAIN INJURY:

In order to be eligible to participate in this study, I must:

* Be between the ages of 18 and 70.
* Have been diagnosed with a TBI by a physician and be at least 6 months post injury
* Have been medically stable for 3 months prior to my most recent TBI.
* Not plan to make any drastic changes to medications (as determined by study staff) for at least 4 weeks.
* Be able to stand unsupported for 5 minutes.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, verbal instructions, and follow-up requirements.

INCLUSION CRITERIA FOR HEALTHY INDIVIDUALS:

In order to be eligible to participate in this study, I must:

* Be between the ages of 18 and 70.
* Not plan to make any drastic changes to medications for at least 4 weeks.
* Not have a history of injury or disease within the last 90 days.
* Be able to stand unsupported for 5 minutes.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, including follow-up requirements.

EXCLUSIONS FOR TRAUMATIC BRAIN INJURY:

I must NOT:

* Have severe cardiac disease such as heart attack or moderate or severe congestive heart failure.
* Have a pre-existing condition resulting in significant disruption in alignment or function of the lower limb during standing.
* Have any additional orthopedic, neuromuscular, or neurological conditions that would interfere with my balance.
* Have had a penetrating TBI (a penetrating TBI is when an item or object goes through the skull to damage the brain).
* Have any previously diagnosed history of balance problems prior to TBI.
* Be able to stand without the ankle foot orthosis (AFO).
* Have fluctuating blood pressure.
* Be on any medication that may affect my balance, strength, or muscle coordination (e.g. Botox).
* Be currently enrolled in another research study that is likely to affect participation in this research study.

EXCLUSIONS FOR HEALTHY INDIVIDUALS:

I must NOT:

* Have a history of injury to my lower limbs in the past 90 days.
* Have severe cardiac disease such as heart attack or moderate or severe congestive heart failure.
* Have a pre-existing condition resulting in significant disruption in alignment or function of the lower limb during standing.
* Have any additional medical conditions that affect my bones, muscles, or nerves that would interfere with my movement or my ability to feel touch or pain.
* Have difficulty following or responding to commands that would limit my study participation.
* Be currently enrolled in another research study that is likely to affect participation in this research study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Assessment | 4 weeks
  A task performance test consisting of 14 items of increasing difficulty graded on a five-point ordinal scale of 0 to 4 (0 = subject is unable to perform task; 4 = subject is independent in performance of task) giving the best possible score of 56 for healthy balance.
Fall Efficacy Scale -International | 4 weeks
  This questionnaire is a widely accepted tool for the assessment of fear of falling and has excellent reliability and validity. It is a self-reported questionnaire that provides information on the level of concern about falls for a range of daily living activities. The original questionnaire contains 16 items and is scored on a four-point scale (1 = not very concerned to 4 = very concerned). Therefore the best possible value is 16 and the worst is 64.
Anticipatory Postural Adjustment- Compensatory Postural Adjustment measures | 4 weeks
  Electromyography 200 ms before the onset of perturbation and 200 ms after the onset of perturbation will be computed for Anticipatory Postural Adjustment- Compensatory Postural Adjustment measures.

SECONDARY OUTCOMES:
Timed up and GO (TUG) | 4 weeks
  TUG is a clinical test of functional gait abilities and dynamic balance. The participants will be asked to walk a distance of 3 meters from a seated position, turn around, walk back to the chair and sit back in the chair.
Center of Mass (CoM) | 4 weeks
  Center of Mass will be collected using Neurocom during small perturbations during quiet standing. All participants will wear a safety harness and a spotter will be present at all times. Root-mean-squared values of CoM displacements will be used for quantifying postural responses.
Center of Pressure (CoP) | 4 weeks
  Center of Pressure will be collected using Neurocom during small perturbations during quiet standing. All participants will wear a safety harness and a spotter will be present at all times. Root-mean-squared values of CoP displacements will be used for quantifying postural responses.
Limits of Stability | 4 weeks
  The limits of stability will be collected using Neurocom. It quantifies the maximum distance the patient can intentionally displace their center of gravity in the four cardinal directions and the four diagonal directions, and maintain stability at those positions.
Joint kinematics | 4 weeks
  Lower extremity joint kinematics (ankle, knee and hip angles) will be computed using Motion Analysis system in the sagittal plane to quantify postural deviations during small perturbations during queit standing using Neurocom. All participants will wear a safety harness and a spotter will be present at all times.
Silver Index | 4 weeks
  Silver index using Movendo Technology platform (Movendo Technology Srl,, Italy) is an objective test that enables to predict falls by assessing static and dynamic balance. Participants will be asked to stand on the Hunova platform. Silver index includes the following tasks: stand with eyes open or eyes closed, stand when the surface is perturbed, move torso on all four sides, perform sit to stand.
Mobility Course | 4 weeks
  Participants will wear Actigraph activity monitor on their wrist, ankle and waist. Their activities (walking in a room about 20 ft long, sitting, standing and walking up and down stairs) will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States